CLINICAL TRIAL: NCT06897423
Title: The Effect of Disaster Midwifery Education Program on Disaster Risk Perception and Self-Efficacy Levels of Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBU-AYDINKARTAL-011
Record Dates: First submitted 2024-12-07; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Disaster Midwifery Training
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (n:40) (Experimental): Midwifery students in the intervention group of the study will receive 8 weeks of disaster midwifery training. The training content will be covered in 8 main categories: "safe prenatal, delivery and postnatal period", "women's reproductive health services", "family planning", "immunization", "violence and sexually transmitted infections" and "newborn and infant care", "reproductive health in disadvantaged groups", "emergency obstetric situations". The training content will be supported by distributing a 12-page training booklet consisting of these contents to the participants. Each training will be planned for 60 minutes.
  Interventions: Other: Education
- Control group (n:40 (No Intervention): no intervention After the research is completed, it is planned to give the same training to the control group.

INTERVENTIONS:
Other: Education — Midwifery students in the intervention group of the study will receive 8 weeks of disaster midwifery training. The training content will be covered in 8 main categories: "safe prenatal, delivery and postnatal period", "women's reproductive health services", "family planning", "immunization", "violence and sexually transmitted infections" and "newborn and infant care", "reproductive health in disadvantaged groups", "emergency obstetric situations".
  Arms: Intervention group (n:40)

SUMMARY:
This research was planned to examine the effect of disaster midwifery education on the disaster risk perception and self-efficacy levels of midwifery students. The research universe will consist of third-year students studying at the Department of Midwifery, Hamidiye Faculty of Health Sciences (HSBF), Health Sciences University (SBU) in the spring semester of the 2023-2024 academic year (N: 80).

In this semi-experimental pre-test and post-test design and control group planned research, in order to determine the sample size; the data were normally distributed, the standard deviation of the main mass was estimated as 1 and the effect size (effect size, difference) as 0.8.

For the analysis to be conducted, it was calculated that the highest power value of the research would be 0.942182 in the case of taking two independent n₁=40, n₂=40 samples at a 5% significance level. The G-power analysis result is given below. Students who volunteer to participate in the study will be assigned to the intervention and control groups using the computer-aided simple random sampling method. Computer-aided randomization will be used in the study, and the number of cases will be entered through the program with the URL address https://www.randomizer.org and random assignment will be made to the intervention and control groups. The study will be conducted single-blind. Midwifery students will be administered the "Disaster Risk Perception" and "Self-Efficacy Scale in Disaster Intervention" before and 8 weeks after the first training. Each training period is limited to 60 minutes, once a week.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research.
* Health Sciences University, Hamidiye Health Sciences Faculty Midwifery Department Being an active student in the 3rd year.

Exclusion Criteria:

* Being a passive student in the 3rd year of the Department of Midwifery, Hamidiye Faculty of Health Sciences, University of Health Sciences.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form: | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, high school graduation, whether they see themselves as sufficient against disasters, etc.
Disaster Risk Perception Scale | 10 minutes
  The scale consists of 21 items and 4 dimensions. The scale has four sub-dimensions: "threat", "fatalism", "controllability" and "anxiety". The "threat" sub-dimension of the scale consists of seven items, the "fatalism" sub-dimension consists of three items, the "controllability" sub-dimension consists of six items and the "anxiety" sub-dimension consists of five items. The items in the scale are in a 5-point Likert format as "1- Strongly Disagree", "2- Disagree", "3-Partially Agree", "4-Agree", "5-Strongly Agree". The lowest score that can be obtained from the scale is 21 and the highest is 105. As the score obtained from the scale increases, the level of disaster risk perception increases.
Self-Efficacy Scale in Disaster Response | 10 minutes
  The Disaster Response Self-Efficacy Scale, developed by Hong-Yan Li and colleagues in 2017 and Turkish validity security studies conducted by Koca and colleagues in 2018, consists of 19 items and 3 sub-dimensions, and the answers are taken with a 5-point Likert scale. A high score from the scale indicates a high level of disaster response self-efficacy. The scale has three sub-factors. Sub-factors: "On-Site Rescue Competence (Items 1 - 11)", "Disaster Psychological Nurse Competence (Items 12 - 15)" and "The nature of the role undertaken in the disaster and adaptation competence (Items 16 - 19)". The Cronbach alpha coefficient for the entire scale is 0.96. The Cronbach alpha values taken for the sub-dimensions are; on-site rescue competence was determined as 0.93, disaster psychological nurse competence was determined as 0.93, the quality of the role undertaken in the disaster and adaptation competence was determined as 0.93

SECONDARY OUTCOMES:
Introductory Information Form: | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, high school graduation, whether they see themselves as sufficient against disasters, etc.
Disaster Risk Perception Scale | 10 minutes
  The scale consists of 21 items and 4 dimensions. The scale has four sub-dimensions: "threat", "fatalism", "controllability" and "anxiety". The "threat" sub-dimension of the scale consists of seven items, the "fatalism" sub-dimension consists of three items, the "controllability" sub-dimension consists of six items and the "anxiety" sub-dimension consists of five items. The items in the scale are in a 5-point Likert format as "1- Strongly Disagree", "2- Disagree", "3-Partially Agree", "4-Agree", "5-Strongly Agree". The lowest score that can be obtained from the scale is 21 and the highest is 105. As the score obtained from the scale increases, the level of disaster risk perception increases.
Self-Efficacy Scale in Disaster Response | 10 minutes
  The Disaster Response Self-Efficacy Scale, developed by Hong-Yan Li and colleagues in 2017 and Turkish validity security studies conducted by Koca and colleagues in 2018, consists of 19 items and 3 sub-dimensions, and the answers are taken with a 5-point Likert scale. A high score from the scale indicates a high level of disaster response self-efficacy. The scale has three sub-factors. Sub-factors: "On-Site Rescue Competence (Items 1 - 11)", "Disaster Psychological Nurse Competence (Items 12 - 15)" and "The nature of the role undertaken in the disaster and adaptation competence (Items 16 - 19)". The Cronbach alpha coefficient for the entire scale is 0.96. The Cronbach alpha values taken for the sub-dimensions are; on-site rescue competence was determined as 0.93, disaster psychological nurse competence was determined as 0.93, the quality of the role undertaken in the disaster and adaptation competence was determined as 0.93

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No